CLINICAL TRIAL: NCT01311375
Title: Evaluation of Omega 3 Supplementation on Neurological Recovery , Lipid Profile and Antioxidant Enzymes and Hormones After Chronic Spinal Cord Injury.
Brief Title: Omega 3 in Intervention Spinal Cord Injured People
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 87-03-85-7538
Record Dates: First submitted 2011-03-06; First posted 2011-03-09 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2012-11

CONDITIONS: Lipid Metabolism Disorders; Peroxidase; Defect
Keywords: spinal,, bone, cord injury, lipid,antioxidant
MeSH Terms: conditions — Lipid Metabolism Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- w3 supplement + capsule CA-D (Experimental): Mor DHA :w3 supp will be given to this group + capsule Ca(500 mg)-D(200 micro gram)
  Interventions: Dietary Supplement: w3 supplement in SCI
- placebo+ CA-D (Placebo Comparator): placebo in the same color,shape,size
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: w3 supplement in SCI — supplements(Mor DHA and Ca "500 mg" -D200 micro g" )( will be given in this group
  Arms: w3 supplement + capsule CA-D
Other: placebo — placebo+ capsule CA-D
  Arms: placebo+ CA-D

SUMMARY:
The objective of this study is to evaluate the effect of omega 3 fatty acid on neurological recovery, lipid profile and Antioxidant system in patients with spinal cord injury. One hundred spinal cord injured patients who come to clinic of spinal injury repair research center selected. Then the patients will receive two supplements capsules of omega 3 (600 mg) in the intervention group and placebo in the control group. Primary outcome measures are professionals evaluation of neurological function by using :

* ASIA scale for sensory and motor function
* FIM scale for Functional potential
* FAM
* SF_36 for quality of life

Lipid profile and Antioxidant profile evaluation by using:

* FBS
* 2hpp
* Insulin
* LDL
* Total cHOL
* TG
* HDL
* Leptin Adiponectin -Calcium-
* 25OHD
* PTH,LH, FSH, Prolactin,Testosterone in males Bone markers by serum levels of :Osteocalcin-Osteoprotegrin_Bone Specified ALP- CTX - RANKL
* BMD

DETAILED DESCRIPTION:
All no neurological evaluation will be done by experiment researcher under considering of a neurologist.All Sub clinical evaluation will be done by specific, sensitive and valid laboratory methods. Intervention time will be 14 months.Comparison of these variables will be done before and after intervention.

ELIGIBILITY:
Inclusion Criteria: no metabolic, malignant or kidney disorder, normal TSH, LH, FSH, prolactin, and testosterone in men and normal prolactin, estradiol, LH, FSH, and TSH in women

Exclusion Criteria:

* pregnancy, lactation, presence of bone disease,hypersensitivity to fish or fish oil, hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-11; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Neurological recovery,metabolic profile and Antioxidant profile evaluation | 4 months
  Primary outcome measures are professionals evaluation of neurological function by using :
  * Osteocalcin
  * osteoprotegrin
  * Bone Specified ALP
  * CTX
  * RANKL
Neurological recovery,metabolic profile and Antioxidant profile evaluation in SCI patients | 14 months
  ASIA scale for sensory and motor function FIM scale for Functional potential FAM
  SF36 for quality of life by using:
  FBS 2hpp Insulin LDL Total cHOL TG HDL Leptin Adiponectin -Calcium- 25OHD PTH,LH, FSH, Prolactin,Testosterone in males

SECONDARY OUTCOMES:
Neurological recovery,metabolic profile and Antioxidant profile evaluation in patients with SCI | 14 months
  BMD : Femur and Lumbar

CONTACTS AND LOCATIONS:
Overall Officials: Abbas Nouroozi, Ph.D, Study Director — Brain and Spinal Cord Injury Repair Research Center
Locations (1):
- Brain and Spinal Injury Repair Research Center, Tehran, Iran